CLINICAL TRIAL: NCT05103228
Title: Cumulative Pregnancy Rate With Lower and Higher Dose of Gonadotropin During Controlled Ovarian Hyperstimulation During IVF Among Expected Poor Responders: a Prospective, Randomized Controlled Trial
Brief Title: Cumulative Pregnancy Rate With Lower and Higher Gonadotropin Dose During IVF Among Poor Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Kovacs MD (Other)
Responsible Party: Sponsor-Investigator, Peter Kovacs MD, Medical Director, Dunamenti REK Istenhegyi IVF Center
Organization: Dunamenti REK Istenhegyi IVF Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52007-13/2021
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Infertility; Ovarian Dysfunction
Keywords: gonadotropin; follitropin alpha; follitropin delta; high-dose gonadotropin; clinical pregnancy; cumulative pregnancy rate
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; follitropin delta; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower gonadotropin dose stimulation (Experimental): Low-dose group:
  * 150 IU follitropin alpha + 75 IU highly purified human menopausal gonadotropin (hpHMG)
  * 10 mcg follitropin delta + 75 IU hpHMG
  Interventions: Drug: Follitropin Alfa; Drug: Follitropin delta; Drug: human menopausal gonadotropin
- Higher gonadotropin dose stimulation (Experimental): High-dose group:
  * 225 IU follitropin alpha + 150 IU highly purified human menopausal gonadotropin (hpHMG)
  * 15 mcg follitropin delta + 150 IU hpHMG
  Interventions: Drug: Follitropin Alfa; Drug: Follitropin delta; Drug: human menopausal gonadotropin

INTERVENTIONS:
Drug: Follitropin Alfa — lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  Other Names: Ovaleap (Theramex Ireland Limited); Bemfola (Richter Gedeon Nyrt., Hungary); Gonal F (Merck Europe B.V.)
Drug: Follitropin delta — lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  Other Names: Rekovelle (Ferring Pharmaceuticals A/S, Denmark)
Drug: human menopausal gonadotropin — lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  Other Names: Menopur (Ferring Pharmaceuticals A/S, Denmark)

SUMMARY:
Controlled ovarian hyperstimulation (COH) is an important step during in vitro fertilization (IVF). Its aim optimally is to recruit 10-15 oocytes. When deciding on the actual treatment, different stimulation protocols, various stimulating agents and wide range of gonadotropin dose can one choose from. Prior to the decision on the actual stimulation protocol and gonadotropin (Gn) dose the patient's expected response to stimulation is assessed primarily using ovarian reserve markers. Most medications used during stimulation exert their effect in a dose-dependent manner hence with a higher Gn dose one would expect a better response, more oocytes. More oocytes could translate into more embryos and potentially a higher pregnancy rate. The currently available evidence however does not support this practice as randomized controlled trials (RCT) have failed to show that the use of higher Gn dose results in higher pregnancy, live-birth rates. These studies however identified patients based on different criteria, compared different stimulation protocols and various Gn doses. There are only two RCTs that compared cumulative live birth rates (fresh + frozen embryo transfers) and they identified poor responders based on different criteria and used different drug regimens. Therefore, the aim of our study is to compare cumulative IVF clinical pregnancy rates using a lower and a higher gonadotropin dose among poor responders identified based on universally accepted criteria.

DETAILED DESCRIPTION:
Background: IVF is started after proper evaluation based on an appropriate indication for the treatment. The first phase of the treatment is the stimulation with the aim to recruit sufficient number of oocytes. In general, 10-15 oocytes are aimed for. This many oocytes should be sufficient for the embryology laboratory procedures and should allow the provider to choose the embryo or embryos for transfer from a larger cohort. More oocytes are associated with more side effects and fewer oocytes limit the efficacy of the laboratory procedures. Stimulation is individualized and usually age, ovarian reserve markers, weight and response to previous stimulation are taken into consideration when decisions are made. Based on ovarian reserve markers patients are grouped as expected normal responders, hyper-responders or poor responders. A poor responder is a patient with low ovarian reserve or low number of oocytes in the ovaries. Their care can be challenging. Different pre-stimulation interventions and various stimulation approaches have been explored in this subset of patients. Typically, providers will prescribe higher gonadotropin doses and expect the retrieval of more oocytes resulting in more transferable embryos. Studies so far however have not supported this practice. In expected poor responders most studies have not shown the collection of more oocytes with higher dose gonadotropins. Those that did find more oocytes described an additional 1-2 oocytes only. None of the studies so far have reported improved pregnancy outcome, including cumulative outcome with more gonadotropins though. The literature is confounded by the various definitions of the poor responder patient, the use of various stimulation protocols in the active treatment versus control groups, the use of oral agents as active treatment and the different clinical endpoints tested (oocyte number, clinical pregnancy, live birth, cumulative live birth). Therefore, we plan to study patients identified as poor responders based on established criteria (POSEIDON criteria). We will use the same stimulation protocols, drug types in the experimental and control groups. We will study clinically meaningful outcomes, live birth rate and cumulative live birth rate.

Design: Investigator initiated prospective, randomized, multi-center, non-blinded trial to compared higher and lower gonadotropin in poor responder patients undegoing IVF-ICSI treatment identified based on Posedion III-IV criteria

Participants: The investigators will enroll patients who, based on their initial evaluation, reproductive history or prior fertility treatment, have a proper indication to undergo in vitro fertilization (IVF)/ intracytoplasmic sperm injection (ICSI) treatment. A basic infertility evaluation includes: 1.) hormonal evaluation of ovarian function, including ovarian reserve testing (anti-Müllerian hormone [AMH] level, antral follicle count [AFC]), 2) transvaginal ultrasound evaluation of female internal genital organs, 3) evaluation of the uterine cavity (hysterosalpingogram, saline sonohysterogram or hysteroscopy), 4) cervical cancer screening, 5) cervical culture for Chlamydia, 6) serologic testing for HIV, hepatitis B, C, syphilis (both partners), 7) semen analysis, 8) male andrological exam, 9) if needed male hormonal +/- genetic testing. IVF-ICSI treatment is started for advanced maternal age, diminished ovarian reserve (DOR), unexplained infertility after failed intrauterine inseminations, male factor infertility, endometriosis.

The investigators plan to recruit:

- infertile patients between the ages of 18-42 who require IVF-ICSI treatment and are identified as poor responders based on: a) AMH: 0.3-1.2 ng/ml or AFC <5, b) AMH>1.2 ng/ml or AFC≥5 but the retrieval of ≤ 4 oocytes during previous IVF treatment. (POSEIDON category III-IV, Alviggi et al. Fertility Sterility 2016)

Methods: prospective, multicenter (5 centers), randomized controlled trial comparing a higher or lower gonadotropin (Gn) dose treatment. In both the low and high groups two different drug regimens (follitropin alpha + hp human menopausal gonadotropin or follitropin delta + hp human menopausal gonadotropin) will be used. 150 IU follitropin alpha was shown to be equally effective to 10 mcg follitropin delta. Therefore, the investigators expect similar response (oocyte yield) with the two regimens within the high and low Gn dose groups but the study design still will allow the investigators to compare the two follitropin medications too, which is a secondary aim.

Lower-dose group:

* 150 IU follitropin alpha + 75 IU highly purified human menopausal gonadotropin (hpHMG)
* 10 mcg follitropin delta + 75 IU hpHMG

Higher-dose group:

* 225 IU follitropin alpha + 150 IU hpHMG
* 15 mcg follitropin delta + 150 IU hpHMG

Treatment protocol:

* The stimulation will get started on day 2 or 3 of the spontaneous menstrual cycle, or on the 5th day after oral contraceptive pill use or after luteal estradiol pretreatment.
* During the stimulation ultrasound +/- serum hormone measurements will be used to monitor response. The first ultrasound is scheduled for day 5 or 6 of stimulation. At the time of the ultrasound blood test for serum estradiol is planned too. At the time of the last scan serum estradiol and progesterone levels will be measured.
* According to the study protocol the patient will continue with the assigned medication dose throughout her treatment. Dose increase is not allowed. If there is evidence for hyper-response [estradiol level > 4000 pmol/l on day 6 or more than 15 follicles over 10 mm any time during the stimulation] the dose can be reduced.
* As soon as two or more follicles reach >17 mm in diameter human chorionic gonadotropin (hCG) or gonadotropin-releasing hormone agonits [GnRH a] trigger injection will be used and 35-36 hours later transvaginal ultrasound guided follicle aspiration will be performed.
* The luteal phase will be supported by vaginal progesterone starting on the day after the retrieval.
* IVF or ICSI fertilization will be performed based on the semen parameters or previous fertilization records.
* The day after the retrieval the success of fertilization will be checked and the embryo(s) will be transferred 2-5 days after the retrieval. Embryo(s) will be transferred transcervically using soft transfer catheters under ultrasound guidance using the afterload technique.
* Surplus good quality embryos will be cryopreserved using vitrification. Elective cryopreservation (no transfer in the fresh cycle) will be performed if: 1) risk of ovarian hyperstimulation syndrome, 2) serum progesterone level over 1.5 ng/ml [5.5 nmol/l] prior to the oocyte collection, 3) any complications between the retrieval and planned fresh transfer (bleeding, infection, illness).
* 12-14 days after the transfer serum human chorionic gonadotropin (HCG) measurement will determine whether implantation has occurred. If the test is positive in 2-3 weeks a vaginal ultrasound will be done to determine the size, location and number of gestational sacs. Viable pregnancies will be referred to a formal prenatal care around week 8-9 of pregnancy. Delivery and perinatal outcome data will be collected by phone call after the delivery.
* If the fresh IVF cycle is not successful but embryos have been cryopreserved then the patient will undergo a frozen embryo transfer treatment cycle either in her own cycle, or in a minimally stimulated or completely artificial cycle.

The care of the patients will not differ from the care of non-study patients in terms of potential medication dose, the number of clinic visits, retrieval and embryology procedures as well as prenatal care.

Randomization: Randomization will be performed according to a computer generated list. (www.randomizer.org) The planned sample size is 700 patients (350 in both the low- and high-dose groups).

Sample size calculation: In order to determine the sample size, the investigators calculated with a 20% pregnancy rate in a patient population that fits the inclusion-exclusion criteria. The investigators expect higher oocyte yield in the higher dose group that should result in more available embryos and therefore more frozen embryo transfers. The investigators calculate that this could increase the cumulative pregnancy rate by 50%. The investigators also believe that about 20% of the patients will drop out for various reasons. Therefore, 350 participants are needed in both arms of the study.

Statistical analysis: After the enrollment of the first 350 patients, a planned interim analysis will be performed to decide whether the planned sample size is sufficient to achieve our goal. Logistic regression analysis using a generalized, mixed linear model will be used to assess the impact of various Gn doses on pregnancy rates. Chi-square test will be used to test significance and OR will be calculated.

Data will be collected for the following parameters:

* Age
* Cycle day 3 follicle stimulating hormone (FSH), estradiol level
* anti-Müllerian hormone (AMH)
* antral follicle count (AFC)
* Indication for IVF: male, tubal, unexplained, endometriosis, diminished ovarian reserve
* Smoking (yes-no)
* Body mass index
* Cycle number (fresh + frozen together)
* Estradiol level on day 6
* Estradiol + progesterone level at the last scan
* Number of follicles >10 mm at the end of stimulation
* Stimulation duration
* Endometrial thickness
* Gn dose (daily, total)
* Trigger mechanism (HCG vs. GnRh agonist)
* Sperm parameters
* Oocyte number
* Mature (MII) oocyte number
* Proportion of mature oocytes (MII/ oocyte number)
* IVF vs. ICSI fertilization
* Number of fertilized (2 pronuclei (PN)) oocytes
* Fertilization rate per oocyte
* Fertilization rate per mature oocyte
* The number of good quality embryos (morphology better than score "6B2" on day 3, or score >2BB on day 5) and proportion of good morphology embryos among all embryos
* Number of transferred embryos
* Number of cryopreserved embryos
* Pregnancy rate (positive hCG)
* Clinical pregnancy rate (sac with viable embryo in it)
* Cumulative pregnancy rate (fresh + frozen embryo transfers)
* Pregnancy/ neonatal outcome

ELIGIBILITY:
Inclusion Criteria:

* Expected poor responder based on:

  1. AMH: 0.3-1.2 ng/ml or AFC <5,
  2. AMH>1.2 ng/ml or AFC≥5 but the retrieval of ≤ 4 oocytes during previous IVF treatment.
* motile sperm with normal morphology obtained from the ejaculate of testicular biopsy
* no more than 3 previous failed IVF cycles (if the patient had 2 or more previous cycles cancelled for poor response she cannot be included)
* BMI: 18-35 kg/m2
* regular 24-35 day cycles
* intact uterine cavity
* indication for in vitro fertilisation treatment (tubal factor, male factor, low ovarian reserve, endometriosis, unexplained infertility)
* age 18-421 yrs

Exclusion Criteria:

* presence of hydrosalpinx
* positive HIV, hepatitis B, C screening tests
* planned preimplantation genetic testing of the embryos
* planned elective cryopreservation
* lack of consent
* not meeting the inclusion criteria

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kovacs, MD, Principal Investigator — Dunamenti REK Istenhegyi IVF Center
Locations (1):
- Dunamenti REK Reprodukciós Központ, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van der Gaast MH, Eijkemans MJ, van der Net JB, de Boer EJ, Burger CW, van Leeuwen FE, Fauser BC, Macklon NS. Optimum number of oocytes for a successful first IVF treatment cycle. Reprod Biomed Online. 2006 Oct;13(4):476-80. doi: 10.1016/s1472-6483(10)60633-5. PMID 17007663
- [Result] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Result] Briggs R, Kovacs G, MacLachlan V, Motteram C, Baker HW. Can you ever collect too many oocytes? Hum Reprod. 2015 Jan;30(1):81-7. doi: 10.1093/humrep/deu272. Epub 2014 Oct 31. PMID 25362088
- [Result] Polyzos NP, Drakopoulos P, Parra J, Pellicer A, Santos-Ribeiro S, Tournaye H, Bosch E, Garcia-Velasco J. Cumulative live birth rates according to the number of oocytes retrieved after the first ovarian stimulation for in vitro fertilization/intracytoplasmic sperm injection: a multicenter multinational analysis including approximately 15,000 women. Fertil Steril. 2018 Sep;110(4):661-670.e1. doi: 10.1016/j.fertnstert.2018.04.039. PMID 30196963
- [Result] Gougeon A. Human ovarian follicular development: from activation of resting follicles to preovulatory maturation. Ann Endocrinol (Paris). 2010 May;71(3):132-43. doi: 10.1016/j.ando.2010.02.021. Epub 2010 Apr 2. PMID 20362973
- [Result] Fleming R, Broekmans F, Calhaz-Jorge C, Dracea L, Alexander H, Nyboe Andersen A, Blockeel C, Jenkins J, Lunenfeld B, Platteau P, Smitz J, de Ziegler D. Can anti-Mullerian hormone concentrations be used to determine gonadotrophin dose and treatment protocol for ovarian stimulation? Reprod Biomed Online. 2013 May;26(5):431-9. doi: 10.1016/j.rbmo.2012.02.027. Epub 2013 Feb 4. PMID 23507133
- [Result] Nelson SM, Yates RW, Lyall H, Jamieson M, Traynor I, Gaudoin M, Mitchell P, Ambrose P, Fleming R. Anti-Mullerian hormone-based approach to controlled ovarian stimulation for assisted conception. Hum Reprod. 2009 Apr;24(4):867-75. doi: 10.1093/humrep/den480. Epub 2009 Jan 10. PMID 19136673
- [Result] Nelson SM. Biomarkers of ovarian response: current and future applications. Fertil Steril. 2013 Mar 15;99(4):963-9. doi: 10.1016/j.fertnstert.2012.11.051. Epub 2013 Jan 8. PMID 23312225
- [Result] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Result] Practice Committee of the American Society for Reproductive Medicine. Electronic address: asrm@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Testing and interpreting measures of ovarian reserve: a committee opinion. Fertil Steril. 2020 Dec;114(6):1151-1157. doi: 10.1016/j.fertnstert.2020.09.134. PMID 33280722
- [Result] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Result] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Result] Leijdekkers JA, Torrance HL, Schouten NE, van Tilborg TC, Oudshoorn SC, Mol BWJ, Eijkemans MJC, Broekmans FJM. Individualized ovarian stimulation in IVF/ICSI treatment: it is time to stop using high FSH doses in predicted low responders. Hum Reprod. 2020 Sep 1;35(9):1954-1963. doi: 10.1093/humrep/dez184. PMID 31838515
- [Result] van Tilborg TC, Torrance HL, Oudshoorn SC, Eijkemans MJC, Koks CAM, Verhoeve HR, Nap AW, Scheffer GJ, Manger AP, Schoot BC, Sluijmer AV, Verhoeff A, Groen H, Laven JSE, Mol BWJ, Broekmans FJM; OPTIMIST study group. Individualized versus standard FSH dosing in women starting IVF/ICSI: an RCT. Part 1: The predicted poor responder. Hum Reprod. 2017 Dec 1;32(12):2496-2505. doi: 10.1093/humrep/dex318. PMID 29121326
- [Result] Liu X, Li T, Wang B, Xiao X, Liang X, Huang R. Mild stimulation protocol vs conventional controlled ovarian stimulation protocol in poor ovarian response patients: a prospective randomized controlled trial. Arch Gynecol Obstet. 2020 May;301(5):1331-1339. doi: 10.1007/s00404-020-05513-6. Epub 2020 Mar 24. PMID 32211953
- [Result] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org. Comparison of pregnancy rates for poor responders using IVF with mild ovarian stimulation versus conventional IVF: a guideline. Fertil Steril. 2018 Jun;109(6):993-999. doi: 10.1016/j.fertnstert.2018.03.019. PMID 29935660
- [Result] Arce JC, Larsson P, Garcia-Velasco JA. Establishing the follitropin delta dose that provides a comparable ovarian response to 150 IU/day follitropin alfa. Reprod Biomed Online. 2020 Oct;41(4):616-622. doi: 10.1016/j.rbmo.2020.07.006. Epub 2020 Jul 15. PMID 32819842
- [Result] Nyboe Andersen A, Nelson SM, Fauser BC, Garcia-Velasco JA, Klein BM, Arce JC; ESTHER-1 study group. Individualized versus conventional ovarian stimulation for in vitro fertilization: a multicenter, randomized, controlled, assessor-blinded, phase 3 noninferiority trial. Fertil Steril. 2017 Feb;107(2):387-396.e4. doi: 10.1016/j.fertnstert.2016.10.033. Epub 2016 Nov 29. PMID 27912901
- [Result] Bosch E, Havelock J, Martin FS, Rasmussen BB, Klein BM, Mannaerts B, Arce JC; ESTHER-2 Study Group. Follitropin delta in repeated ovarian stimulation for IVF: a controlled, assessor-blind Phase 3 safety trial. Reprod Biomed Online. 2019 Feb;38(2):195-205. doi: 10.1016/j.rbmo.2018.10.012. Epub 2018 Dec 14. PMID 30594482
- [Result] Ishihara O, Klein BM, Arce JC; Japanese Follitropin Delta Phase 2 Trial Group. Randomized, assessor-blind, antimullerian hormone-stratified, dose-response trial in Japanese in vitro fertilization/intracytoplasmic sperm injection patients undergoing controlled ovarian stimulation with follitropin delta. Fertil Steril. 2021 Jun;115(6):1478-1486. doi: 10.1016/j.fertnstert.2020.10.059. Epub 2020 Dec 4. PMID 33272623

RESULTS

PARTICIPANT FLOW:
Groups:
- Lower Gonadotropin Dose Stimulation: Low-dose group:
  * 150 IU follitropin alpha + 75 IU highly purified human menopausal gonadotropin (hpHMG)
  * 10 mcg follitropin delta + 75 IU hpHMG
  Follitropin Alfa: lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  Follitropin delta: lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  human menopausal gonadotropin: lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
- Higher Gonadotropin Dose Stimulation: High-dose group:
  * 225 IU follitropin alpha + 150 IU highly purified human menopausal gonadotropin (hpHMG)
  * 15 mcg follitropin delta + 150 IU hpHMG
  Follitropin Alfa: lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  Follitropin delta: lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
  human menopausal gonadotropin: lower dose gonadotropin (follitropin alpha/ follitropin delta + hpHMG) vs. higher dose stimulation (Follitropin alpha/delta + hpHMG)
Period: Overall Study
Arm/Group | Lower Gonadotropin Dose Stimulation | Higher Gonadotropin Dose Stimulation
Started | 98 | 92
Completed | 94 | 91
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Gonadotropin Dose Stimulation | Higher Gonadotropin Dose Stimulation | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (3.3) | 37.1 (3.6) | 37.0 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 91 | 185
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Anti-Müllerian hormone [Mean (Standard Deviation); unit: ng/ml] | 0.7 (0.3) | 0.7 (0.2) | 0.7 (0.2)
Antral follicle count [Mean (Standard Deviation); unit: piece] | 5.8 (2.5) | 6.0 (2.5) | 6.0 (2.0)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.8 (4.4) | 24.1 (4.1) | 23.8 (4.6)
Cycle number [Mean (Standard Deviation); unit: cycles] | 1.8 (1.1) | 1.7 (1.0) | 1.7 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Clinical Pregnancy Rate
Description: an ultrasound confirmation of an intrauterine gestational sac with an embryo with detectable heartbeat in it after the fresh + if available frozen embryo transfer treatments
Time Frame: 18 months
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Gonadotropin Dose Stimulation | Higher Gonadotropin Dose Stimulation
Number analyzed (Participants) | 94 | 91
Participants | 27 | 17

2. Secondary Outcome: Live Birth Rate
Description: delivery of a viable newborn after 24 weeks gestation
Time Frame: 12 months
Population: Intentition to treat population
Measure: Number; unit: live births
Arm/Group | Lower Gonadotropin Dose Stimulation | Higher Gonadotropin Dose Stimulation
Number analyzed (Participants) | 94 | 91
live births | 15 | 10

3. Secondary Outcome: Cumulative Live Birth Rate
Description: Cumulative live birth: delivery of a viable newborn after 24 weeks gestation after the fresh embryo transfer or if it is unsuccessful but surplus embryos were frozen then after any of the subsequent frozen embryo transfer cycles. All these transfers (fresh and frozen) are the result of a single stimulation. If a live birth is reached during the fresh or any of the subsequent frozen transfers from the same stimulation then it is considered a positive outcome; if the fresh transfer or any of the subsequent frozen transfers from the same stimulation do not result in a live birth it is considered a negative result.
Time Frame: 12 months
Measure: Number; unit: live births
Arm/Group | Lower Gonadotropin Dose Stimulation | Higher Gonadotropin Dose Stimulation
Number analyzed (Participants) | 94 | 91
live births | 17 | 13

ADVERSE EVENTS:
Time Frame: 4 weeks if the pregnancy test is negative: from start of the study drug administration up to the pregnancy test. 8 weeks if the pregnancy test is positive: from start of the study drug administration up to the first ultrasound confirming the pregnancy.
Description: SAE were colected for based on standard definitions.
Arm/Group | Lower Gonadotropin Dose Stimulation | Higher Gonadotropin Dose Stimulation
All-Cause Mortality (participants affected / at risk) | 0/94 | 1/91
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/91
Other Adverse Events (participants affected / at risk) | 0/94 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT05103228/Prot_SAP_000.pdf